CLINICAL TRIAL: NCT05497843
Title: An Open-label, Multicenter, Phase II Study of Chiauranib Capsule in Patients With Advanced or Unresectable Soft Tissue Sarcoma Previously Failed to Standard of Care Treatment
Brief Title: Chiauranib for Advanced or Unresectable Soft Tissue Sarcoma(STS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAR204; NCT05542433 (obsolete NCT alias)
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — chiauranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chiauranib capsule (Experimental): Patients take chiauranib capsules 50mg, orally once daily, 21 days as a cycle until objective disease progression
  Interventions: Drug: Chiauranib

INTERVENTIONS:
Drug: Chiauranib — 50mg, orally once daily
  Other Names: CS2164

SUMMARY:
This is a Phase 2, single-arm, open-label study in patients with advanced or unresectable soft tissue sarcoma.

DETAILED DESCRIPTION:
This single-arm, open-label, multiple-center clinical trial aims to study the efficacy and safety of chiauranib in the treatment of patients with advanced or unresectable soft tissue sarcoma, and to explore potential biomarkers associated with chiauranib, as well as their correlation and clinical benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years and ≤75 years.
2. Histologically confirmed advanced or unresectable soft tissue sarcoma with failure of standard therapy or no standard therapy.
3. At least one measurable target lesion as defined by RECIST1.1, i.e., a lesion that has radiologic evidence of disease progression, after treatment with radiotherapy or local-regional therapy
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
5. Laboratory criteria are as follows:

   1. Hematology: absolute neutrophil count (ANC) ≥1.5×109/L, platelet ≥75×109/L, hemoglobin ≥80 g/L.
   2. Biochemistry: serum creatinine <1.5×upper limit of normal (ULN), total bilirubin ≤1.5×ULN, both alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (≤5×ULN for patients with hepatic metastasis).
   3. Coagulation panel: international normalized ratio (INR) <1.5.
6. Life expectancy of at least 3 months.
7. Willingness to sign a written informed consent document.

Exclusion Criteria:

1. Active central nervous system (CNS) symptoms during the screening period and/or CNS metastases requiring hormone therapy within 28 days before the first dose, or lesions involving the brain stem or pia mater.
2. Imaging during the screening period showed that the tumor had invaded the periphery of the important blood vessels or the investigator judged that the tumor was likely to invade the important blood vessels and cause massive bleeding during the trial.
3. Pleural fluid, ascites or pericardial effusion with significant symptoms or required treatment of puncture or drainage during the screening period.
4. Current or previous history of other malignancies (other than adequately treated basal or squamous cell carcinoma of the skin or cervical carcinoma in situ) unless curative treatment has been performed and there is no evidence of recurrence or metastasis in the last 5 years
5. Prior treatment with vascular endothelial growth factor(VEGF)/vascular endothelial growth factor receptor(VEGFR) inhibitor, like Apatinib, Anlotinib, Fruquintinib, Bevacizumab, etc., or Aurora kinase inhibitors (For patients eligible for anlotinib, only those who could not receive anlotinib for various reasons were allowed to be enrolled in this study. Patients who had previously received anlotinib were excluded from the study).
6. Anti-tumor treatments such as radiotherapy, chemotherapy, immunotherapy and targeted therapy were used within 28 days before the first treatment.
7. Allergic or contraindicated to any component or vehicle of the test drug.
8. Treatment with an investigational agent/instrument within 28 days prior to first dose.
9. Prior major surgery or trauma within 28 days prior to first dose and/or presence of any non-healing wound, fracture, or ulcer during the screening period.
10. Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1(except alopecia) during the screening period.
11. Uncontrolled or significant cardiovascular disease, including:

    1. New York Heart Association (NYHA) class II or higher congestive heart failure, unstable angina pectoris, myocardial infarction occurred within 6 months before the first dose, or an arrhythmia requiring treatment during the screening period with a left ventricular ejection fraction (LVEF) of <50%.
    2. Primary cardiomyopathy (dilated cardiomyopathy, hypertrophic cardiomyocyte, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy).
    3. Clinically significant history of QTc interval prolongation, or screening QTc interval >470ms for women and >450ms for men.
    4. Symptomatic coronary heart disease requiring medical treatment during the screening period.
    5. Records of concomitant use of ≥3 antihypertensive drug components within 14 days prior to the first dose, or systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg during the screening period (at rest, approximately 5 minutes apart, three consecutive measurements, averaged).
    6. Previous hypertensive crisis or hypertensive encephalopathy.
    7. Other condition investigator considered inappropriate.
12. Chest imaging during the screening period revealed interstitial lung disease or pulmonary fibrosis or pulmonary inflammation requiring treatment, or a history of pneumonia treated with oral or intravenous steroids within 6 months before the first dose.
13. Significant gastrointestinal abnormalities during the screening period that were judged by the investigator to be likely to interfere with drug intake, transport, or absorption (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, post-small bowel resection, etc.), or total gastrectomy, or a history of gastrointestinal perforation and/or fistula within 6 months prior to the first dose.
14. 24-hour urine protein quantitative examination must be performed when urine protein ≥2+ in routine urine examination during the screening period. Patients cannot be enrolled if quantitative urine protein ≥ 1g/24 h.
15. Active bleeding within 2 months before the first dose, or taking anticoagulants during the screening period (e.g., warfarin, phenprocoumon, and allow prophylactic use of low-dose aspirin and low-molecular weight heparin), Or investigator judged that there was a high risk of bleeding during the screening period (such as esophageal and gastric fundus varices with bleeding risk, locally active ulcer lesions, positive fecal occult blood could not exclude gastrointestinal bleeding, intermittent hemoptysis, etc.).
16. A history of deep vein thrombosis or pulmonary embolism or a thrombotic event such as a cerebrovascular accident within 6 months before the first dose (implantable venous port or catheter-derived thrombosis, investigator evaluation for enrollment).
17. Active infections that required systemic treatment during the screening period (oral, intravenous infusion).
18. HIV antibody positive during the screening period.
19. hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive with virus replication, hepatitis C antibody (HCV-Ab) positive with virus replication during the screening period.
20. Any mental or cognitive impairment that may limit the understanding, execution, and adherence to the study.
21. Drug use and long-term alcohol abuse affected the evaluation of test results.
22. Pregnant or lactating women; Be unwilling or unable to during the treatment of this test and test the last 12 weeks after the treatment using effective methods of contraception among women of reproductive age [women of childbearing age include: did not receive any had menstruation and successful artificial sterilization (hysterectomy and bilateral tubal ligation or bilateral oophorectomy) or menstruating]; If the partner is a woman of childbearing age, the subject is a fertile man who is not using effective contraception.
23. Other conditions considered by the investigator to be inappropriate for trial participation, such as concomitant disease, concomitant therapy, or any laboratory abnormality, may interfere with the evaluation of efficacy and safety results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival of 12 weeks(PFS12w) | 12 weeks after the first dose
  Proportion of subjects who did not have disease progression or recurrence (according to RECIST1.1) or death from any cause at week 12 after receiving medical treatment

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  Proportion of participants who have a partial response (PR) or complete response (CR) to therapy according to RECIST 1.1
Progression-free survival (PFS) | Up to 2 years
  From the first time of treatment until the date of first documented progression or date of death from any cause, whichever comes first
Duration of response (DOR) | Up to 2 years
  From the first date of response until the date of first documented progression
Disease control rate (DCR) | Up to 2 years
  Proportion of participants in partial, complete or stable disease according to RECIST 1.1.
Overall survival (OS) | Up to 2 years
  From the first dose of treatment until the date of death from any cause
Safety and Tolerability | Up to 28 days after the last dose
  Incidence of adverse events (AEs) as assessed by CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xing Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No